CLINICAL TRIAL: NCT06867705
Title: Digital Monitoring With Patient-Reported Outcomes in Cancer Care: A Randomized Controlled Trial RC - 102 (Resilience Care - 102)
Brief Title: Randomized Controlled Trial of Remote Symptoms Monitoring With Resilience PRO Compared to Care As Usual Only
Acronym: RC-102
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Resilience (Industry)
Collaborators: UNICANCER (Other); Sanoia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-102; 2024-A01584-43 (ID RCB) (Other: Agence Nationale de Sécurité du Médicament (ANSM)); N° Eudamed: CIV-25-01-050834 (Other: Agence Nationale de Sécurité du Médicament (ANSM))
Record Dates: First submitted 2025-02-21; First posted 2025-03-10 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Remote Patient Monitoring; Remote Symptom Monitoring; Digital medicine; Resilience PRO; Resilience; PRO; Patient-reported Outcomes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote Symptoms Monitoring with Resilience PRO (Experimental): Resilience PRO will be added on top of conventional care
  Interventions: Device: Resilience PRO
- Usual care without Remote Symptoms Monitoring (No Intervention): Conventional care only

INTERVENTIONS:
Device: Resilience PRO — The patient will use Resilience PRO remote symptoms monitoring.
  Arms: Remote Symptoms Monitoring with Resilience PRO

SUMMARY:
The goal of this clinical trial is to learn if Resilience PRO, a digital solution performing remote symptoms monitoring, can improve the quality of life of patients with a diagnosis of cancer receiving systemic anticancer treatment.

The main question it aims to answer is:

- Do patients with a diagnosis of cancer receiving systemic anticancer therapy and using Resilience PRO have an improved quality of life? Researchers will compare patients using Resilience PRO plus care as usual to patients receiving care as usual only.

Participants in the intervention arm will use Resilience PRO, a mobile phone application regularly asking participants about their symptoms. For clinically important symptoms, an alert is sent to the care team that can incorporate that information to timely adjust the care of the participants. Participants both in the control arm and in the intervention arm will further receive care as usual.

DETAILED DESCRIPTION:
Resilience PRO is a digital medical device (dMD CE marked, class IIa) that enables the remote monitoring of patients diagnosed with cancer receiving anticancer systemic therapy. Resilience PRO has been positively evaluated by the French health authorities (HAS, Haute Autorité de Santé) and is registered on the French LATM list (Liste des Activités de Télésurveillance Médicale).

Resilience PRO is a software medical device prescribed by cancer treating physicians to collect electronic patient-reported outcomes (ePRO). The Resilience PRO workflow comprises the following steps:

* Step 1. Collection of ePRO
* Step 2. Intelligent analysis and alerts
* Step 3. Adapted care

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults ≥ 18 years.
* Informed Consent: Patient giving signed informed consent to participate in the RC - 102 clinical study.
* Diagnosis: Patients with cancer at any stage.
* Systemic Treatment
* Remote Monitoring Eligibility: Access to a smartphone
* Language: Ability to understand and communicate in the language(s) in which the trial is conducted.

Exclusion Criteria:

* Age: Patients under 18 years of age.
* Life Expectancy: Patients with a life expectancy of less than 6 months as estimated by the treating physician.
* Concurrent remote monitoring
* HSCT or CAR-T Therapy
* Cognitive Impairment
* Pregnancy or breastfeeding
* Subject under administrative or judicial control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1458 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Health-Related quality of life | 3 months
  EORTC QLQ-C30

SECONDARY OUTCOMES:
Health-economic evaluation | 12 months
  The outcome is measured in QALYs. These are calculated from the EQ-5D-5L questionnaire scores.
Overall survival | 36 months

OTHER OUTCOMES:
Experience from patients | 12 months
  Patient experience and usability of the RPM system survey (Patient-Reported Experience Measures PREMs)
Experience from HCP | 12 months
  Healthcare Professionals Experience survey.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Scotté, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (28):
- France (26):
  - Hôpital Privé de Provence, Aix-en-Provence
  - Centre Hospitalier du Pays d'Aix - Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence
  - Centre Hospitalier Henri Mondor-Aurillac, Aurillac
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Centre Hospitalier Universitaire de Caen Normandie, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire Grenoble - Alpes, La Tronche
  - GHICL Hôpital Saint Vincent de Paul, Lille
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital Privé Jean Mermoz - Institut de Cancérologie, Lyon
  - AP-HM Assistance Publique - Hôpitaux de Marseille Hôpital de la Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hôpital Privé du Confluent, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - AP-HP Hôpitaux Universitaires La Pitié Salpêtrière, Paris
  - Clinique Mutualiste Bretagne Occidentale, Quimper
  - Hôpital Privé de la Loire (HPL) - Saint Etienne, Saint-Etienne
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Centre Hospitalier Universitaire Sud Réunion, Saint-Pierre
  - Centre Clinical Elsan, Soyaux
  - Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer, Toulon
  - Clinique Pasteur, Toulouse
  - Centre de Cancérologie Les Dentellières, Valenciennes
  - Clinique Teissier, Valenciennes
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsklinikum Schleswig-Holstein (UKSH), Campus Kiel, Kiel
  - Universitätsklinikum Schleswig-Holstein (UKSH), Campus Lübeck, Lübeck

REFERENCES:
- See also: EUDAMED - European Database on Medical Devices — https://ec.europa.eu/tools/eudamed/#/screen/search-device/4295460b-cbc2-49a2-8f50-cb1d9dbf2453